CLINICAL TRIAL: NCT06930495
Title: The Effect of Adiposity on Muscle and Microvascular Function in HFpEF
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Hearon, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0279
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: HFpEF; Weight loss; adiposity; inflammation; RNA sequencing; skeletal muscle
MeSH Terms: conditions — Weight Loss; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFpEF and Obesity Group: Patients with HFpEF (heart failure with preserved ejection fraction) and diabetes will undergo standard of care treatment using the most appropriate second-generation anti-diabetic drug that induces clinically significant weight loss after completing baseline (pre) testing.
  Interventions: Drug: Weight loss SOC Treatment with second generation anti-diabetic medications
- Control Group (Non-HFpEF and Obesity): Controls matched for age and hypertension

INTERVENTIONS:
Drug: Weight loss SOC Treatment with second generation anti-diabetic medications — To determine the best incretin-based drug for the treatment [done as part of regular standard of care (SOC) treatment], participants will go to UTSW weight wellness clinic and undergo a comprehensive history and physical exam to evaluate their overall health. This information is used to create an individualized approach to the participants weight loss regimen. As part of the regimen, participants will receive guidance on initiating lifestyle modifications including diet and exercise and may be referred to a clinical psychologist for evaluation and management of factors like stress, anxiety and depression, and exercise which may influence their health behaviors and body weight.
  Groups: HFpEF and Obesity Group

SUMMARY:
This project is an observational study in patients with heart failure with preserved ejection fraction (HFpEF) who are candidates for treatment with weight loss medication to manage obesity or diabetes as part of their standard clinical care. This study will include multiple experimental visits before and after treatment (minimum 7 percent weight loss, between 9-12 months) to understand how increased adiposity and inflammation effects skeletal muscle and cardiovascular health and function and to examine the effect of medically directed weight loss on skeletal muscle health and exercise tolerance.

The objective of this study is to

1. Define the mechanisms by which adiposity impairs exercise hemodynamics, microvascular function, and oxygen transport/utilization in patients with HFpEF.
2. Determine if intensive medically directed weight loss can reduce microvascular inflammation and normalize exercise hemodynamics.
3. Quantify the effect of medically directed weight loss on skeletal muscle function and catabolism.

Hypotheses

1. Perfusion of subcutaneous adipose tissue disrupts blood flow distribution and impairs muscle microvascular perfusion and exercise hemodynamics.
2. Extramyocellular muscular lipid deposition and microvascular endothelial inflammation is associated with reduced capillarity and impaired microvascular perfusions, while intramyocellular triglyceride content is associated with poor skeletal muscle oxidative capacity,
3. Intensive weight loss will improve exercise hemodynamics, microvascular perfusion, and reduce muscular inflammation, and resistance training will augment these effects.

DETAILED DESCRIPTION:
Objective one will also include a cross-sectional comparison between HFpEF patients before treatment and non-HFpEF controls matched for age and hypertension

ELIGIBILITY:
Inclusion Criteria:

Group 1: Patients with HFpEF

* Diagnosis of heart failure or clear heart failure hospitalization
* Stable ejection fraction > 0.50
* Objective evidence of elevated left ventricular filling pressure by one of the following i) pulmonary capillary wedge pressure ≥25 mmHg during supine cardiopulmonary exercise testing or ii) a change in pulmonary capillary wedge pressure of >15 mmHg during upright exercise
* Must be candidates for pharmacological incretin-based directed intensive weight loss therapies as part of their SOC
* BMI>32kg/m2
* ≥45 years old
* Incretin naïve for 6 months

Group 2: Non-HFpEF controls

* Adults who do not have heart failure with preserved ejection fraction
* Age ≥ 18 years

Exclusion Criteria:

Group 1

* Prior history of reduced ejection fraction (<50%)
* Infiltrative cardiomyopathy
* NYHA Class IV chronic heart failure
* Left bundle branch block
* Unstable coronary artery disease
* Uncontrolled arrhythmia
* CKD 4 or higher
* Currently taking incretin-based drugs (SGL2, GLP1)
* Severe valvular heart disease
* BMI > 50kg/m2
* Other debilitating illness that would preclude participation
* Any contra-indication to MRI
* Any contra-indication to muscle biopsies.

Group 2

* Age < 18 years
* BMI > 50 kg/m2
* Atrial fibrillation with poorly controlled heart rate
* PDE5 inhibitor use
* Severe valvular disease
* Severe COPD
* CKD 4 or higher
* Currently taking incretin-based drugs (SGL2, GLP1)
* Any contra-indication to MRI
* Any contra-indication to muscle biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with HFpEF
  - UTSW HFpEF clinic: lead by Dr. Ambarish Pandey
  Group 2: non-HFpEF controls
  * subjects in the UTSW volunteer research registry who meet inclusion/exclusion criteria
  * community outreach (emailers, word of mouth, referrals)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak muscle perfusion during exercise | Pre intervention (Day 1)
  Peak muscle perfusion (Aβ) during exercise will be assessed by Contrast enhanced ultrasound (CEU)
Peak muscle perfusion during exercise | Post intervention (Post Day 1)
  Peak muscle perfusion (Aβ) during exercise will be assessed by Contrast enhanced ultrasound (CEU)
Single cell RNA sequencing of skeletal muscle | Pre intervention (Day 2)
  Skeletal muscle biopsies will be taken from the vastus lateralis using the modified Bergstrom technique and immediately prepared for single cell RNA sequencing. Samples will be digested, filtered, washed and resuspended in freezing media and checked for concentration and viability before single cell RNA sequencing is performed
Single cell RNA sequencing of skeletal muscle | Post intervention (Day 2)
  Skeletal muscle biopsies will be taken from the vastus lateralis using the modified Bergstrom technique and immediately prepared for single cell RNA sequencing. Samples will be digested, filtered, washed and resuspended in freezing media and checked for concentration and viability before single cell RNA sequencing is performed
Muscle to fat ratio of leg | Pre intervention (Day 3)
  MRI of the leg will be performed to acquire clear visualization of fasciae separating different muscle groups and thus allowing for quantification of intermuscular fat (muscle:fat ratio)
Peak change in microvascular perfusion from rest to exercise | Pre intervention (Day 3)
  MRI of the leg will be performed utilizing the PIVOT sequence which will measure global and regional perfusion of blood to the muscles in the lower leg at rest and during exercise. the peak change will be reported as the change from baseline to peak exercise
Muscle to fat ratio of leg | Post intervention (Day 3)
  MRI of the leg will be performed utilizing the PIVOT sequence which will measure the change in perfusion of blood to the muscles in the lower leg from rest to during exercise
Peak change in microvascular perfusion from rest to exercise | Post intervention (Day 3)
  MRI of the leg will be performed utilizing the PIVOT sequence which will measure global and regional perfusion of blood to the muscles in the lower leg at rest and during exercise. the peak change will be reported as the change from baseline to peak exercise

SECONDARY OUTCOMES:
Vascular function - endothelium dependent vasodilation | Pre intervention (Day1)
  A small ultrasound probe will be placed over the brachial artery and a small blood pressure cuff will be positioned on the lower arm, just below the elbow. Images of the vessel will be continuously recorded for 1 min (baseline) before the cuff is inflated to a high pressure (220mmHg) for 5minutes and immediately after the cuff is deflated for 3 minutes. The change in brachial artery diameter following deflation of cuff from baseline will represent a marker of vascular function
Vascular function - endothelium dependent vasodilation | Post intervention (Day 1)
  A small ultrasound probe will be placed over the brachial artery and a small blood pressure cuff will be positioned on the lower arm, just below the elbow. Images of the vessel will be continuously recorded for 1 min (baseline) before the cuff is inflated to a high pressure (220mmHg) for 5minutes and immediately after the cuff is deflated for 3 minutes. The change in brachial artery diameter following deflation of cuff from baseline will represent a marker of vascular function
Blood volume measurement | Pre intervention (Day1)
  The carbon monoxide rebreathe technique will be performed to measure blood volume
Blood volume measurement | Post intervention (Day 1)
  The carbon monoxide rebreathe technique will be performed to measure blood volume
2min walk endurance test | Pre intervention (Day 2)
  Participants will be asked to walk on a flat surface back and forth between 2 cones for 2minutes. the total distance covered (in meters) during the 2-minutes will be recorded as a marker of endurance
Hand grip strength | Pre intervention (Day 2)
  Participants will squeeze a handheld dynamometer as hard as they can to measure handgrip strength (in kg). This will be performed on both hands
2min walk endurance test | Post intervention (Day2)
  Participants will be asked to walk on a flat surface back and forth between 2 cones for 2minutes. the total distance covered (in meters) during the 2-minutes will be recorded as a marker of endurance
Hand grip strength | Post intervention (Day2)
  Participants will squeeze a handheld dynamometer as hard as they can to measure handgrip strength (in kg). This will be performed on both hands
Body composition | Pre intervention (Day 0)
  measured using dual xray absorptiometry (DEXA) to get lean mass, muscle mass, body fat percentage
Body composition | Post intervention (Day 1)
  measured using dual xray absorptiometry (DEXA) to get lean mass, muscle mass, body fat percentage
Apnea hypopnea index | Pre intervention (Day 2)
  Participants will be given an at home sleep apnea test that is incorporated into a wrist-based wearable that enables non-invasive tracking of sleep apnea burden.
  Sleep apnea will be determined from the apnea hypopnea index measured by the device. Apnea hypopnea index will be calculated as the average number of apneas or hypopneas that occurs per hour of sleep
Apnea hypopnea index | Post intervention (Day 2)
  Participants will be given an at home sleep apnea test that is incorporated into a wrist-based wearable that enables non-invasive tracking of sleep apnea burden.
  Sleep apnea will be determined from the apnea hypopnea index measured by the device. Apnea hypopnea index will be calculated as the average number of apneas or hypopneas that occurs per hour of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Hearon Jr, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No